CLINICAL TRIAL: NCT01681212
Title: Phase 2 Study of Ipilimumab Plus Dacarbazine in Japanese Patients With Previously Untreated Unresectable or Metastatic Melanoma
Brief Title: Phase 2 Study of Ipilimumab Plus Dacarbazine in Japanese Patients With Advanced Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA184-202
Record Dates: First submitted 2012-09-05; First posted 2012-09-07 (Estimated); Results first posted 2015-06-11 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-06

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ipilimumab, 10 mg/kg + Dacarbazine, 850 mg/m^2 (Experimental): During the Induction Period, participants received ipilimumab, 10 mg/kg, as tolerated by intravenous (IV) infusion as 1 single dose during Weeks 1 (Day 1), 4, 7, and 10 for a total of 4 separate doses. During the Maintenance Phase, participants received ipilimumab, 10 mg/kg, as tolerated by IV infusion every 12 weeks, beginning at Week 24, until disease progression or unacceptable toxicity occurred or the patient withdrew consent. Participants also received dacarbazine, 850 mg/m^2, by IV infusion over 30 to 60 minutes, starting on Week 1 and repeated every 3 weeks until Week 22. Dacarbazine was dosed on the same day as ipilimumab, when applicable, after the ipilimumab dose.
  Interventions: Drug: Ipilimumab; Drug: Dacarbazine

INTERVENTIONS:
Drug: Ipilimumab
  Other Names: BMS-734016
Drug: Dacarbazine

SUMMARY:
The purpose of this study is to determine the survival rate after 1 year of treatment with ipilimumab plus dacarbazine in patients with previously untreated Stage III (unresectable) or Stage IV melanoma.

ELIGIBILITY:
Key inclusion criteria:

* Japanese patients with histologic diagnosis of malignant melanoma
* Previously untreated Stage III with N3 (unresectable) or Stage IV melanoma
* Prior adjuvant melanoma therapy permitted
* Eastern Cooperative Oncology Group performance status of 0 or 1
* Life expectancy of at least 16 weeks in this study
* Adequate bone marrow and renal and hepatic function, specifically:

  * white blood cell count ≥2500/uL, absolute neutrophil count ≥1000/uL, platelet count ≥75,000/uL, hemoglobin level ≥9.0 g/dL, creatinine level ≤2.5*upper limit of normal (ULN), aspartate transaminase/alanine transaminase level <2.5*ULN for patients without liver metastasis and <5*ULN for patients with liver metastasis, total bilirubin level <1.5*ULN (for those with Gilbert's Syndrome, lower than 3.0 mg/dL)

Key exclusion criteria:

* Evidence of brain metastases on brain imaging
* Active brain metastases with symptoms or requiring corticosteroid treatment; patients with any other malignancy from which they have been disease-free for fewer than 5 years, with the exception of adequately treated and cured basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix
* Primary ocular or mucosal melanoma
* History of or current active autoimmune disease
* History or concurrent disease of gastrointestinal perforations
* HIV infection; active Hepatitis B or C or human T-lymphotropic virus type1 infection, based on testing performed during the screening period of this study
* Prior or concomitant therapy with any anticancer agent for melanoma, or other investigational anticancer therapies
* Prior adjuvant therapy <4 weeks prior to the start of study drug administration
* Concomitant therapy with immunosuppressive agents, surgery, or radiotherapy
* Prior treatment with CTLA-4 inhibitors/agonists or other experimental immunotherapy drugs
* Treatment with other investigational products within 4 weeks prior to initial treatment of study drug

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (6):
- Japan (6):
  - Local Institution, Fukuoka, Fukuoka
  - Local Institution, Kumamoto, Kumamoto
  - Local Institution, Matsumoto-shi, Nagano
  - Local Institution, Sunto-gun, Shizuoka
  - Local Institution, Chuo-ku, Tokyo
  - Local Institution, Chuo-shi, Yamanashi

REFERENCES:
- [Derived] Yamazaki N, Uhara H, Fukushima S, Uchi H, Shibagaki N, Kiyohara Y, Tsutsumida A, Namikawa K, Okuyama R, Otsuka Y, Tokudome T. Phase II study of the immune-checkpoint inhibitor ipilimumab plus dacarbazine in Japanese patients with previously untreated, unresectable or metastatic melanoma. Cancer Chemother Pharmacol. 2015 Nov;76(5):969-75. doi: 10.1007/s00280-015-2870-0. Epub 2015 Sep 25. PMID 26407818
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 21 participants were enrolled, and 15 received treatment.
Groups:
- Ipilimumab, 10 mg/kg + Dacarbazine, 850 mg/m^2: During the Induction Period, participants received ipilimumab, 10 mg/kg, as tolerated by intravenous (IV) infusion as 1 single dose during Weeks 1 (Day 1), 4, 7, and 10 for a total of 4 separate doses. During the Maintenance Phase, participants received ipilimumab, 10 mg/kg, as tolerated by IV infusion every 12 weeks, beginning at Week 24, until disease progression, unacceptable toxicity, or withdrawal of consent. Participants also received dacarbazine, 850 mg/m^2, by IV infusion over 30 to 60 minutes, starting on Week 1 and repeated every 3 weeks until Week 22. Dacarbazine was dosed on the same day as ipilimumab, when applicable, after the ipilimumab dose.
Period: Overall Study
Arm/Group | Ipilimumab, 10 mg/kg + Dacarbazine, 850 mg/m^2
Started | 21 (Enrolled)
Received Treatment | 15
Completed | 15 (Completed=patients who received treatment; not completed=patients who did not receive treatment)
Not Completed | 6
Not completed — No longer met study criteria | 5
Not completed — Administrative reason by sponsor | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of treatment medication
Arm/Group | Ipilimumab, 10 mg/kg + Dacarbazine, 850 mg/m^2
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.0 (12.66)
Age, Customized [Number; unit: Participants]
  Younger than 65 | 10
  65 and older | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Race/Ethnicity, Customized [Number; unit: Participants]
  Japanese | 15
  Other | 0
Female Age, Continuous [Mean (Standard Deviation); unit: Years] — Data are provided for the 5 women in the study.
  Years | 47.2 (13.26)
M-stage at study entry [Number; unit: Participants] — M-stage=stage of metastases (M), based on criteria of the American Joint Committee on Cancer. M1A=metastases to skin, subcutaneous tissue, or distant lymph nodes. M1B=metastases to lung. M1C=metastases to all other visceral sites or distant metastases to any site combined with an elevated serum level of lactase dehydrogenase.
  Participants
    M0 | 1
    M1B | 7
    M1C | 7
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: Participants] — ECOG scales are used to assess the progress of disease and the disease's effects on daily living abilities and to determine appropriate treatment. Grade 0=fully active; able to carry on all activities without restriction. Grade 1=restricted in strenuous activity but ambulatory; able to perform light work. Grade 2=ambulatory; capable of all self care but unable to work; up more than 50% of waking hours. Grade 3=capable of limited self care, confined to bed or chair more than 50% of waking hours. Grade 4=Completely disabled; cannot carry on any self care; totally confined to bed or chair.
  Participants
    0 | 13
    1 | 2
Height [Mean (Standard Deviation); unit: Centimeters] | 163.0 (9.28)
Female age, customized [Number; unit: Participants] — Data are provided for the 5 women in the study.
  Participants
    Younger than 50 years | 3
    50 years and older | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Surviving at 1 Year
Description: Survival rate=percentage of participants surviving at 1 year following start of study drug. Every effort was made to collect survival data on all patients, including those withdrawn from treatment for any reason. If the death of a patient was not reported, the patient's last known alive date was recorded. Confidence intervals were computed using the Clopper-Pearson method.
Time Frame: At 1 year from start of study drug
Population: All participants who received at least 1 dose of study drug.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Ipilimumab, 10 mg/kg + Dacarbazine, 850 mg/m^2
Number analyzed (Participants) | 15
Percentage of participants | 66.7 [42.3 to 85.8]

2. Secondary Outcome: Number of Participants With Grade 3-4 Immune-related Adverse Events (irAEs)
Description: irAEs are adverse events of unknown cause, consistent with an immune phenomenon, and considered to be causally related to drug exposure. Six subcategories of irAE are assessed: gastrointestinal, liver, skin, endocrine, neurologic, and other. The irAEs are programmatically determined from a predefined list of MedDRA terms. irAEs will be measured every 3 weeks in induction phase, every 6 weeks in Maintenance Phase to Week 48, and every 12 weeks until Progressive Disease. Grading criteria: Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe, Grade 4=Life-threatening or disabling, Grade 5=Death.
Time Frame: First dose to 90 days following last dose of study drug
Population: All participants who received at least 1 dose of study drug
Measure: Number; unit: Participants
Arm/Group | Ipilimumab, 10 mg/kg + Dacarbazine, 850 mg/m^2
Number analyzed (Participants) | 15
Participants
  All Grade 3-4 irAEs | 11
  Skin irAEs | 10
  Liver irAEs | 12
  Gastrointestinal irAEs | 6
  Endocrine irAEs | 3
  Neurologic irAEs | 0
  Other irAEs | 2

3. Secondary Outcome: Number of Patients Who Died and Who Had Serious Adverse Events (SAEs), Treatment-related SAEs, Adverse Events (AEs) Leading to Discontinuation, Related AEs Leading to Discontinuation, Related AEs, Grade 3-4 AEs, and Related Grade 3-4 AEs
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Related=having certain, probable, possible, or unknown relationship to study drug. Grade 1=mild; Grade 2=moderate; Grade 3=severe; Grade 4=life-threatening or disabling; Grade 5=death.
Time Frame: First dose to 90 days following last dose of study drug. All deaths were poststudy, occurring more than 90 days after the last dose of study drug.
Population: All participants who received at least 1 dose of study drug
Measure: Number; unit: Participants
Arm/Group | Ipilimumab, 10 mg/kg + Dacarbazine, 850 mg/m^2
Number analyzed (Participants) | 15
Participants
  Deaths | 5
  SAEs | 14
  Related SAEs | 11
  AEs leading to discontinuation | 9
  Related AEs leading to discontinuation | 9
  AEs Grade 3-4 | 11
  Related AEs | 15
  Related Grade 3-4 AEs | 11

ADVERSE EVENTS:
Arm/Group | Ipilimumab, 10 mg/kg + Dacarbazine, 850 mg/m^2
Serious Adverse Events (participants affected / at risk) | 14/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimumab, 10 mg/kg + Dacarbazine, 850 mg/m^2 (N=15)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Alanine aminotransferase increased (Investigations) | 10
Back pain (Musculoskeletal and connective tissue disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Aspartate aminotransferase increased (Investigations) | 7
Dizziness (Nervous system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimumab, 10 mg/kg + Dacarbazine, 850 mg/m^2 (N=15)
Blood thyroid stimulating hormone increased (Investigations) | 2
Constipation (Gastrointestinal disorders) | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Electrocardiogram ST-T change (Investigations) | 1
Headache (Nervous system disorders) | 1
Malaise (General disorders) | 2
Oral herpes (Infections and infestations) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Bone marrow failure (Blood and lymphatic system disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Flushing (Vascular disorders) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 3
Influenza like illness (General disorders) | 2
Lymph node pain (Blood and lymphatic system disorders) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1
Ulcer (General disorders) | 1
Weight increased (Investigations) | 1
Alanine aminotransferase increased (Investigations) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 3
Gastritis (Gastrointestinal disorders) | 1
Mucosal inflammation (General disorders) | 1
Oedema peripheral (General disorders) | 2
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Radiation skin injury (Injury, poisoning and procedural complications) | 1
Sinusitis (Infections and infestations) | 1
Vascular pain (Vascular disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Cushingoid (Endocrine disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 3
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 5
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Fungal infection (Infections and infestations) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Nasopharyngitis (Infections and infestations) | 1
Nausea (Gastrointestinal disorders) | 7
Splenomegaly (Blood and lymphatic system disorders) | 1
Weight decreased (Investigations) | 4
Abdominal pain upper (Gastrointestinal disorders) | 1
Aspartate aminotransferase increased (Investigations) | 7
Blood lactate dehydrogenase increased (Investigations) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 3
Insomnia (Psychiatric disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 1
Pyrexia (General disorders) | 4
Vision blurred (Eye disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2
Chest pain (General disorders) | 1
Eosinophil count increased (Investigations) | 1
Fatigue (General disorders) | 1
Gamma-glutamyltransferase increased (Investigations) | 2
Hepatic steatosis (Hepatobiliary disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypophysitis (Endocrine disorders) | 1
Injection site pain (General disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Phlebitis (Vascular disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 2
Herpes zoster (Infections and infestations) | 1
Oedema (General disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 6
Amylase increased (Investigations) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2
Extravasation (General disorders) | 1
Folliculitis (Infections and infestations) | 1
Hepatomegaly (Hepatobiliary disorders) | 2
Hypothyroidism (Endocrine disorders) | 2
Pneumonia (Infections and infestations) | 1
Presyncope (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 2
Tinea pedis (Infections and infestations) | 1

LIMITATIONS AND CAVEATS:
This study was discontinued due to severe liver toxicity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.